CLINICAL TRIAL: NCT06749418
Title: Role of the Mineralocorticoid Receptor in Microvascular Endothelial Dysfunction After Preeclampsia
Brief Title: Vascular Effects of High-Salt After Preeclampsia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202408643
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Preeclampsia; Preeclampsia Postpartum
MeSH Terms: conditions — Pre-Eclampsia | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- High-salt supplement (Experimental): Participants will be counseled to consume a low-salt diet (<2000 mg/day of sodium) for 10 days. After 3 days of a low-salt diet, participants will consume the high-salt supplement (4500 mg/day) for 7 days while maintaining a low-salt diet. On days 3 and 10, participants will arrive at the laboratory where the investigators will assess microvascular endothelial function. Blood will be collected to investigate circulating angiotensin II responses to low- (day 3) and high- (day 10) salt diet. On days 2 and 9, participants will undergo ambulatory blood pressure monitoring and 24-hour urine collection.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Local heating: eplerenone is locally and acutely delivered to the cutaneous microvasculature during local heating of the skin to assess endothelium-dependent dilation, L-NAME is added to assess nitric oxide-dependent dilation during this response.

SUMMARY:
Women who develop preeclampsia during pregnancy are more likely to develop and die of cardiovascular disease later in life, even if they are otherwise healthy. Importantly, women who had preeclampsia have an exaggerated vascular responsiveness to hypertensive stimuli, such as high-salt intake, compared to women who had a healthy pregnancy. The reason why this occurs is unclear but may be related to impaired endothelial function and dysregulation of the angiotensin system that occurs during the preeclamptic pregnancy and persists postpartum, despite the remission of clinical symptoms. While the association between a history of preeclampsia and vascular dysfunction leading to elevated CVD risk is well known, the mechanisms underlying this dysfunction remains unclear.

The purpose of this study is to examine the role of vascular mineralocorticoid receptor, the terminal receptor in the angiotensin system that contributes to blood pressure regulation, in mediating exaggerated microvascular endothelial dysfunction before and after a high-salt stimulus. This will help us better understand the mechanisms of microvascular dysfunction these women, and how inhibition of these receptors may improve microvascular function.

In this study, we use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) we examine the blood vessels in a nickel-sized area of the skin.

ELIGIBILITY:
Inclusion Criteria:

* women who had preeclampsia and women who did not have preeclampsia
* 12 weeks to 5 years postpartum
* 18-45 years old

Exclusion Criteria:

* history of hypertension or metabolic disease before pregnancy
* history of gestational diabetes
* history of gestational hypertension without preeclampsia
* skin diseases
* current tobacco use
* current antihypertensive medication
* statin or other cholesterol-lowering medication
* currently pregnant
* body mass index less than 18.5 kg/m2
* allergy to materials used during the experiment.(e.g. latex),
* known allergy to study drugs or salt-supplement

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in microvascular endothelial function following local eplerenone treatment compared to placebo treatment measured by laser-Doppler flowmetry | Day 3 (low-salt diet run in) and Day 10 (low-salt diet + high-salt supplement)
  Cutaneous vascular vasodilator response (cutaneous conductance; %max) to local heating of the skin; intradermal microdialysis for the local delivery of eplerenone compared to control (Ringer's solution), followed by L-NAME infusion to quantify NO-dependent response
Changes in 24-hour urine sodium | Day 2, Day 9
  The investigators will measure urine sodium to ensure differences in salt-take between low- and high-salt.

SECONDARY OUTCOMES:
Changes in circulating aldosterone concentrations | Day 3, Day 10
  The investigators will collect blood at the start of each experiment to determine differences in aldosterone concentrations between low- and high-salt.
Changes in circulating angiotensin II concentrations | Day 3, Day 10
  The investigators will collect blood at the start of each experiment to determine differences in circulating angiotensin II concentrations between low- and high-salt.
Changes in ambulatory blood pressure | Day 2, Day 9
  The investigators will measure ambulatory blood pressure, assessed as mean arterial pressure calculated from measured systolic and diastolic pressures, responses to low- and high-salt.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Reid-Stanhewicz, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No